CLINICAL TRIAL: NCT04408066
Title: Specimen Collection for Development and Performance Evaluation of the LumiraDx Platform Point of Care Tests for Sars-Cov-2 IgG/IgM & Antigen to be Used as an Aid in Diagnosis of COVID-19
Brief Title: COVID-19: A POC Test Under Research & Evaluation
Acronym: CAPTURE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Number of required participants met
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00028
Record Dates: First submitted 2020-04-30; First posted 2020-05-29 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
Keywords: POC; IVD; SARS-CoV-2; IgG; IgM; Antigen; Antibody
MeSH Terms: conditions — COVID-19 | interventions — Specimen Handling

STUDY DESIGN:
Intervention Model Description: A Sample Collection & Performance Evaluation Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A:Suspected COVID-19 patients (Experimental): Arm A: Suspected COVID-19 Patients - SARS-CoV-2 viral antigen test swab and blood sample for SARS-CoV-2 IgG/IgM
  Interventions: Diagnostic Test: Sample Collection/Performance Evaluation (A)
- Arm B: Previously positive COVID-19 patients (Experimental): Arm B: Previously Positive COVID-19 patients - SARS-CoV-2 IgG/IgM blood sample. Capillary fingerstick samples will additionally be collected in Stage 2.
  Interventions: Diagnostic Test: Sample Collection/Performance Evaluation (B)

INTERVENTIONS:
Diagnostic Test: Sample Collection/Performance Evaluation (A) — This is a prospective sample collection and performance evaluation study which involves no therapeutic intervention.
  Sample types include:
  * Nasal/Throat/Nasal Throat Combo/ Nasopharyngeal (as per sites SOC) Swab
  * Whole Venous Blood
  Arms: Arm A:Suspected COVID-19 patients
Diagnostic Test: Sample Collection/Performance Evaluation (B) — This is a prospective sample collection and performance evaluation study which involves no therapeutic intervention.
  Sample types include:
  * Whole Venous Blood
  * Fingerstick Capillary Sample
  Arms: Arm B: Previously positive COVID-19 patients

SUMMARY:
Collection of nasal/nasopharyngeal/throat swabs and blood samples from patients presenting at their designated care facility displaying symptoms of COVID-19 and undergoing a SOC SARS-CoV-2 test or those who have tested positive in the past to aid development, calibration and performance evaluation for the LumiraDx POC test.

DETAILED DESCRIPTION:
CAPTURE is a two-stage sample collection study to complete the development, calibration and performance evaluation phases of the LumiraDx Point of Care (POC) device for the detection of the SARS-CoV-2 virus and the SARS-CoV-2 IgG/IgM status of infected patients. The study is split into two arms targeting separate populations throughout each stage.

Stage 1: Consists of sample collection only, to facilitate the in-house development and calibration of the LumiraDx SARS-CoV-2 assays.

Stage 2: Consists of sample collection to facilitate the performance evaluation of the LumiraDx SARS-CoV-2 studies. In this stage the testing will be completed onsite using the LumiraDx POC device.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years of age.
2. Patient meets either of the below categories:

   1. Patient is presenting with symptoms indicative of COVID-19 and will be completing SOC sampling for SARS-CoV-2 PCR testing. (Eligible for Arm A)
   2. Patient has had a confirmed positive SARS-CoV-2 PCR test result in the past. (Eligible for Arm B)

Exclusion Criteria:

1. The patient does not have the capacity to consent as determined by the Research Team (and the impartial witness if applicable).
2. The patient is deemed to be unsuitable for research at the research teams' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the LumiraDx Assay versus reference methods with regards to clinical sensitivity and specificity for the detection of the SARS-COV-2 IgG/IgM and viral antigen in patient samples. | 1 Year approx
  Primary Outcome - To collect sufficient SARS-CoV-2 samples (nasal/nasopharyngeal/throat swabs and blood samples) to aid development, calibration and performance evaluation of the LumiraDx POC test. Results will be used to asses performance of the LumiraDx assay versus reference methods with regards to the clinical sensitivity and specificity for the detection of the SARS-COV-2 IgG/IgM and viral antigen in patient samples.

CONTACTS AND LOCATIONS:
Overall Officials: Samer Elkhodair, Principal Investigator — University College London Hospitals
Locations (3):
- United Kingdom (3):
  - Barts Health NHS Trust, London
  - Homerton University Hospital NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No